CLINICAL TRIAL: NCT01811758
Title: Culturally Specific Interventions and Acculturation in African American Smokers
Brief Title: Culturally Specific Interventions: African American Smokers
Acronym: SB2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Monica W. Hooper, Associate Professor, University of Miami
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SmokeBreak2
Record Dates: First submitted 2013-03-12; First posted 2013-03-15 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Smoking; Smoking Cessation
Keywords: Culturally Specific Cognitive Behavioral Therapy; Standard Cognitive Behavioral Therapy
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Culturally Specific CBT (Experimental): Culturally specific cognitive behavioral therapy. Group format, 8 sessions, approximately 90 minutes. Up to 8-weeks of transdermal nicotine patches. Focused on African Americans: smoking patterns, health outcomes, discrimination, stress, weight concerns, cultural beliefs and practices.
  Interventions: Behavioral: Culturally Specific CBT
- Standard CBT (control) (Active Comparator): Standard cognitive behavioral therapy. Group format, 8 sessions, approximately 90 minutes each. Up to 8-weeks of transdermal nicotine patches. Traditional CBT, with no focus on race: smoking and health, benefits of quitting, weight control, relapse prevention, coping skills.
  Interventions: Behavioral: Standard CBT

INTERVENTIONS:
Behavioral: Culturally Specific CBT
  Arms: Culturally Specific CBT
Behavioral: Standard CBT
  Arms: Standard CBT (control)

SUMMARY:
The investigators expect that a culturally specific group intervention targeting African American smokers will result in greater smoking cessation rates compared to a standard intervention.

ELIGIBILITY:
Inclusion Criteria:

1. self-identification as African American
2. current smoker of ≥ 5 cigarettes/day or expired CO level of ≥ 8 ppm;
3. age 18-65;
4. able to speak and read English;
5. permanent contact information;
6. access to transportation by public transit or car;
7. no current behavioral or pharmacological treatment ;
8. interest in quitting smoking; (9) have availability to attend sessions.

Exclusion Criteria:

1. enrolled in another cessation program,
2. do not speak and read English,
3. do not have access to transportation by car or bus to attend sessions,
4. do not have childcare during session times,
5. have contraindications for patch use (pregnant/breastfeeding),
6. if they are in treatment for substance abuse (e.g., illicit drugs, alcohol abuse),
7. if they endorse active addiction to another substance (e.g., illicit drugs or alcohol),
8. if they have been diagnosed with an acute cardiac or respiratory condition;
9. people identified as having a severe mental illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence | Overall effect at 12-months
  Generalized linear mixed model of overall intervention effect.

SECONDARY OUTCOMES:
7-day point prevalence abstinence | 6-months

CONTACTS AND LOCATIONS:
Overall Officials: Monica Hooper, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

REFERENCES:
- [Background] Hooper MW, Larry R, Okuyemi K, Resnicow K, Dietz NA, Robinson RG, Antoni MH. Culturally specific versus standard group cognitive behavioral therapy for smoking cessation among African Americans: an RCT protocol. BMC Psychol. 2013 Aug 21;1(1):15. doi: 10.1186/2050-7283-1-15. eCollection 2013. PMID 25566367